CLINICAL TRIAL: NCT07294989
Title: Median Effective Concentration of Ciprofol and Its Correlation With Bispectral Index: A Prospective Observational Study
Brief Title: The Effective Blood Concentration of Ciprofol
Status: Recruiting | Type: Observational
Sponsor: Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-117
Record Dates: First submitted 2025-06-25; First posted 2025-12-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Disease
MeSH Terms: conditions — Thyroid Diseases | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ciprofol group: Anesthesia induction was achieved through target-controlled infusion of ciprofol.
  Interventions: Drug: Ciprofol

INTERVENTIONS:
Drug: Ciprofol — Beginning with an initial target plasma concentration of ciprofol at 1.2 μg/mL. Assessments of the Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scale and Bispectral Index (BIS) values are performed every minute until the patient achieves a complete anesthetic state (defined as an MOAA/S score of 0).

SUMMARY:
1. Eligible patients were selected and enrolled in the study.
2. General anesthesia was induced using ciprofol in all participants, with standardized evaluation of consciousness levels during induction.
3. The patients' pain and cognition are followed up after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Scheduled for elective thyroidectomy
* ASA physical status classification I-II
* Willing to participate and providing written informed consent

Exclusion Criteria:

* Recent use of sedatives or opioid analgesics
* Severe hepatic or renal dysfunction defined as:Child-Pugh class C (score ≥10), Creatinine clearance <35 mL/min ,Requiring preoperative dialysis
* Significant cardiovascular comorbidities
* Body mass index ≥35 kg/m² or <18.5 kg/m²
* Known hypersensitivity or adverse reactions to propofol/ciprofol
* Neuropsychiatric disorders including:Alzheimer's disease,History of cerebrovascular events,Traumatic brain injury,Space-occupying brain lesions,Other significant neurological deficits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective thyroidectomy at Peking University Shenzhen Hospital
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The effect-site concentration of cipofol, when MOAAS reaches 2 | From the beginning of anesthesia induction until 1 minute after intubation, the MOAA/S score was assessed every minute, with simultaneous recording of the effect-site concentration (Ce).
  The effect-site concentration of cipofol corresponding to MOAA/S score (Modified Observer's Assessment of Alertness/Sedation) of 2.
  (Modified Observer's Assessment of Alertness/Sedation: 5--Responds readily to name spoken in normal tone ； 4--Lethargic response to name spoken in normal tone ； 3--Responds only after name is called loudly and/or repeatedly ； 2--Responds only after mild prodding or shaking ；
  1--Responds only after painful trapezius squeeze ； 0--No response after painful trapezius squeeze；)

SECONDARY OUTCOMES:
The effect-site concentration of cipofol, when MOAA/S reaches 0. | From the beginning of anesthesia induction until 1 minute after intubation, the MOAA/S score was assessed every minute, with simultaneous recording of the effect-site concentration (Ce).
  The effect-site concentration of cipofol corresponding to MOAA/S score (Modified Observer's Assessment of Alertness/Sedation) of 0.
Bispectral index | From the beginning of anesthesia induction until 1 minute after intubation, the MOAA/S score was assessed every minute, with simultaneous recording of the BIS values.
  Bispectral Index (BIS) values corresponding to different Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scores.
The EC₅₀ and EC₉₅ of ciprofol | From the beginning of anesthesia induction until 1 minute after intubation , the MOAA/S score was assessed every minute, with simultaneous recording of the effect-site concentration (Ce).
  The EC₅₀ and EC₉₅ of ciprofol corresponding to MOAA/S scores of 2 and 0
Heart rate | From the beginning of anesthesia induction until 1 minute after intubation, the MOAA/S score was assessed every minute, with simultaneous recording of the HR.
  Heart rate(in bpm) corresponding to different Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scores.
Blood pressure | From the beginning of anesthesia induction until 1 minute after intubation, the MOAA/S score was assessed every minute, with simultaneous recording of the systolic blood pressure, diastolic blood pressure and mean arterial pressure.
  The systolic blood pressure, diastolic blood pressure and mean arterial pressure corresponding to different MOAAS scores were all recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

REFERENCES:
- [Background] Glen JB. The development of 'Diprifusor': a TCI system for propofol. Anaesthesia. 1998 Apr;53 Suppl 1:13-21. doi: 10.1111/j.1365-2044.1998.53s115.x. PMID 9640110
- [Background] Shafer SL, Gregg KM. Algorithms to rapidly achieve and maintain stable drug concentrations at the site of drug effect with a computer-controlled infusion pump. J Pharmacokinet Biopharm. 1992 Apr;20(2):147-69. doi: 10.1007/BF01070999. PMID 1629794
- [Background] Absalom AR, Glen JI, Zwart GJ, Schnider TW, Struys MM. Target-Controlled Infusion: A Mature Technology. Anesth Analg. 2016 Jan;122(1):70-8. doi: 10.1213/ANE.0000000000001009. PMID 26516798
- [Background] Zbinden AM, Maggiorini M, Petersen-Felix S, Lauber R, Thomson DA, Minder CE. Anesthetic depth defined using multiple noxious stimuli during isoflurane/oxygen anesthesia. I. Motor reactions. Anesthesiology. 1994 Feb;80(2):253-60. doi: 10.1097/00000542-199402000-00004. PMID 8311307
- [Background] Smith C, McEwan AI, Jhaveri R, Wilkinson M, Goodman D, Smith LR, Canada AT, Glass PS. The interaction of fentanyl on the Cp50 of propofol for loss of consciousness and skin incision. Anesthesiology. 1994 Oct;81(4):820-8; discussion 26A. PMID 7943832
- [Background] Eger EI 2nd, Saidman LJ, Brandstater B. Minimum alveolar anesthetic concentration: a standard of anesthetic potency. Anesthesiology. 1965 Nov-Dec;26(6):756-63. doi: 10.1097/00000542-196511000-00010. No abstract available. PMID 5844267
- [Background] Gu Y, Hao J, Wang J, Liang P, Peng X, Qin X, Zhang Y, He D. Effectiveness Assessment of Bispectral Index Monitoring Compared with Conventional Monitoring in General Anesthesia: A Systematic Review and Meta-Analysis. Anesthesiol Res Pract. 2024 Aug 7;2024:5555481. doi: 10.1155/2024/5555481. eCollection 2024. PMID 39149130
- [Background] Chiang MH, Wu SC, Hsu SW, Chin JC. Bispectral Index and non-Bispectral Index anesthetic protocols on postoperative recovery outcomes. Minerva Anestesiol. 2018 Feb;84(2):216-228. doi: 10.23736/S0375-9393.17.12033-X. Epub 2017 Oct 12. PMID 29027770
- [Background] Rosow C, Manberg PJ. Bispectral index monitoring. Anesthesiol Clin North Am. 2001 Dec;19(4):947-66, xi. doi: 10.1016/s0889-8537(01)80018-3. PMID 11778388
- [Result] Guo X, Qiao Y, Yin S, Luo F, Yi L, Chen J, Lu M. Pharmacokinetics and pharmacodynamics of ciprofol after continuous infusion in elderly patients. BMC Anesthesiol. 2025 Jan 27;25(1):41. doi: 10.1186/s12871-025-02907-4. PMID 39871139
- [Result] Liu L, Wang K, Yang Y, Hu M, Chen M, Liu X, Yan P, Wu N, Xiang X. Population pharmacokinetic/pharmacodynamic modeling and exposure-response analysis of ciprofol in the induction and maintenance of general anesthesia in patients undergoing elective surgery: A prospective dose optimization study. J Clin Anesth. 2024 Feb;92:111317. doi: 10.1016/j.jclinane.2023.111317. Epub 2023 Nov 15. PMID 37976683
- [Result] Irwin MG, Hui TW, Milne SE, Kenny GN. Propofol effective concentration 50 and its relationship to bispectral index. Anaesthesia. 2002 Mar;57(3):242-8. doi: 10.1046/j.0003-2409.2001.02446.x. PMID 11879213
- [Result] Kateliya R, Madhukant, Dubey M, Chandra S, Sahay N. Comparison of recovery profiles in target-controlled infusions (TCI) versus manually controlled infusions for total intravenous anesthesia (TIVA) in laparoscopic surgeries. A randomized controlled trial. J Anaesthesiol Clin Pharmacol. 2023 Apr-Jun;39(2):258-263. doi: 10.4103/joacp.joacp_396_21. Epub 2023 Apr 19. PMID 37564857
- [Result] Mu J, Jiang T, Xu XB, Yuen VM, Irwin MG. Comparison of target-controlled infusion and manual infusion for propofol anaesthesia in children. Br J Anaesth. 2018 May;120(5):1049-1055. doi: 10.1016/j.bja.2017.11.102. Epub 2018 Feb 3. PMID 29661382
- [Result] Hu C, Horstman DJ, Shafer SL. Variability of target-controlled infusion is less than the variability after bolus injection. Anesthesiology. 2005 Mar;102(3):639-45. doi: 10.1097/00000542-200503000-00024. PMID 15731604
- [Result] Russell D, Wilkes MP, Hunter SC, Glen JB, Hutton P, Kenny GN. Manual compared with target-controlled infusion of propofol. Br J Anaesth. 1995 Nov;75(5):562-6. doi: 10.1093/bja/75.5.562. PMID 7577281
- [Result] Nimmo AF, Absalom AR, Bagshaw O, Biswas A, Cook TM, Costello A, Grimes S, Mulvey D, Shinde S, Whitehouse T, Wiles MD. Guidelines for the safe practice of total intravenous anaesthesia (TIVA): Joint Guidelines from the Association of Anaesthetists and the Society for Intravenous Anaesthesia. Anaesthesia. 2019 Feb;74(2):211-224. doi: 10.1111/anae.14428. Epub 2018 Oct 31. PMID 30378102
- [Result] Perez-Otal B, Aragon-Benedi C, Pascual-Bellosta A, Ortega-Lucea S, Martinez-Ubieto J, Ramirez-Rodriguez JM; Research Group in Anaesthesia, Resuscitation, and Perioperative Medicine of Institute for Health Research Aragon (ISS Aragon). Neuromonitoring depth of anesthesia and its association with postoperative delirium. Sci Rep. 2022 Jul 26;12(1):12703. doi: 10.1038/s41598-022-16466-y. PMID 35882875
- [Result] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Result] Daccache N, Wu Y, Jeffries SD, Zako J, Harutyunyan R, Pelletier ED, Laferriere-Langlois P, Hemmerling TM. Safety and recovery profile of patients after inhalational anaesthesia versus target-controlled or manual total intravenous anaesthesia: a systematic review and meta-analysis of randomised controlled trials. Br J Anaesth. 2025 May;134(5):1474-1485. doi: 10.1016/j.bja.2025.02.007. Epub 2025 Mar 11. PMID 40074622
- [Result] Yang D, Zhou J, Sun L, Li M, Zhang J. Comparison of postoperative awakening between ciprofol and propofol in elderly patients undergoing hip replacement surgery: a single-blind, randomized, controlled trial. Minerva Anestesiol. 2024 Dec;90(12):1074-1081. doi: 10.23736/S0375-9393.24.18263-6. Epub 2024 Dec 3. PMID 39625705
- [Result] Chen L, Xie Y, Du X, Qin W, Huang L, Dai J, Qin K, Huang J. The Effect of Different Doses of Ciprofol in Patients with Painless Gastrointestinal Endoscopy. Drug Des Devel Ther. 2023 Jun 12;17:1733-1740. doi: 10.2147/DDDT.S414166. eCollection 2023. PMID 37333965
- [Result] Li J, Wang X, Liu J, Wang X, Li X, Wang Y, Ouyang W, Li J, Yao S, Zhu Z, Guo Q, Yu Y, Meng J, Zuo Y. Comparison of ciprofol (HSK3486) versus propofol for the induction of deep sedation during gastroscopy and colonoscopy procedures: A multi-centre, non-inferiority, randomized, controlled phase 3 clinical trial. Basic Clin Pharmacol Toxicol. 2022 Aug;131(2):138-148. doi: 10.1111/bcpt.13761. Epub 2022 Jun 10. PMID 35653554
- [Result] Teng Y, Ou M, Wang X, Zhang W, Liu X, Liang Y, Li K, Wang Y, Ouyang W, Weng H, Li J, Yao S, Meng J, Shangguan W, Zuo Y, Zhu T, Liu B, Liu J. Efficacy and safety of ciprofol for the sedation/anesthesia in patients undergoing colonoscopy: Phase IIa and IIb multi-center clinical trials. Eur J Pharm Sci. 2021 Sep 1;164:105904. doi: 10.1016/j.ejps.2021.105904. Epub 2021 Jun 8. PMID 34116176
- [Result] Teng Y, Ou MC, Wang X, Zhang WS, Liu X, Liang Y, Zuo YX, Zhu T, Liu B, Liu J. Pharmacokinetic and pharmacodynamic properties of ciprofol emulsion in Chinese subjects: a single center, open-label, single-arm dose-escalation phase 1 study. Am J Transl Res. 2021 Dec 15;13(12):13791-13802. eCollection 2021. PMID 35035718
- [Result] Hu C, Ou X, Teng Y, Shu S, Wang Y, Zhu X, Kang Y, Miao J. Sedation Effects Produced by a Ciprofol Initial Infusion or Bolus Dose Followed by Continuous Maintenance Infusion in Healthy Subjects: A Phase 1 Trial. Adv Ther. 2021 Nov;38(11):5484-5500. doi: 10.1007/s12325-021-01914-4. Epub 2021 Sep 24. PMID 34559359
- [Result] Liao J, Li M, Huang C, Yu Y, Chen Y, Gan J, Xiao J, Xiang G, Ding X, Jiang R, Li P, Yang M. Pharmacodynamics and Pharmacokinetics of HSK3486, a Novel 2,6-Disubstituted Phenol Derivative as a General Anesthetic. Front Pharmacol. 2022 Feb 3;13:830791. doi: 10.3389/fphar.2022.830791. eCollection 2022. PMID 35185584
- [Result] de Gasperi A, Mazza E, Noe L, Corti A, Cristalli A, Prosperi M, Sabbadini D, Savi MC, Vai S. Pharmacokinetic profile of the induction dose of propofol in chronic renal failure patients undergoing renal transplantation. Minerva Anestesiol. 1996 Jan-Feb;62(1-2):25-31. PMID 8768021
- [Result] Bian Y, Zhang H, Ma S, Jiao Y, Yan P, Liu X, Ma S, Xiong Y, Gu Z, Yu Z, Huang C, Miao L. Mass balance, pharmacokinetics and pharmacodynamics of intravenous HSK3486, a novel anaesthetic, administered to healthy subjects. Br J Clin Pharmacol. 2021 Jan;87(1):93-105. doi: 10.1111/bcp.14363. Epub 2020 Aug 3. PMID 32415708
- [Result] Petkar S, Bele A, Priya V, Bawiskar D. Pharmacological Insights and Clinical Applications of Ciprofol: A Narrative Review. Cureus. 2024 Aug 28;16(8):e68034. doi: 10.7759/cureus.68034. eCollection 2024 Aug. PMID 39347129
- [Result] Curro JM, Santonocito C, Merola F, Messina S, Sanfilippo M, Brancati S, Drago F, Sanfilippo F. Ciprofol as compared to propofol for sedation and general anesthesia: a systematic review of randomized controlled trials. J Anesth Analg Crit Care. 2024 Apr 8;4(1):24. doi: 10.1186/s44158-024-00159-1. PMID 38589912
- [Result] He KQ, Huang TT, Tan MY, Gao C, Wang S. Efficacy and Safety of Ciprofol Versus Propofol as Anesthetic for Patients Undergoing Painless Colonoscopy. Pain Ther. 2024 Dec;13(6):1633-1644. doi: 10.1007/s40122-024-00662-x. Epub 2024 Oct 14. PMID 39400664